CLINICAL TRIAL: NCT06803082
Title: The Impact of Systemic Light Chain Amyloidosis on Eyes and Its Appendages
Brief Title: The Impact of Systemic Light Chain Amyloidosis on Eyes
Acronym: Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KYPJ080; 82322016 (Other Grant/Funding Number: National Natural Science Foundation of China Outstanding Young Scientists Fund Program)
Record Dates: First submitted 2024-12-13; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-08

CONDITIONS: Systemic Light Chain Amyloidosis; Ocular Complications
Keywords: Systemic Light Chain Amyloidosis; Ocular Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Exposed group: Ocular Complications of Systemic Light Chain Amyloidosis. Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
- Unexposed group: Unexposed group: patients without Systemic Light Chain Amyloidosis

SUMMARY:
Study Purpose and Principle: Amyloidosis is a group of diseases characterized by the deposition of amyloid proteins in tissues and organs throughout the body, with common affected organs including kidneys, heart, nervous system, gastrointestinal tract, and liver. Nowadays, nearly 40 different proteins have been found to form amyloid fibrils in body, among which Systemic Light Chain (AL) Amyloidosis is the most common type of systemic amyloidosis. AL amyloidosis is a plasma cell disorder, with its precursor protein originating from free light chains produced by abnormal plasma cell clones, which form amyloid substances that deposit in tissues and organs causing lesions. In terms of incidence, the incidence of AL amyloidosis is 8-10 cases per million person-years in the United States and is considered a rare disease in our country. AL amyloidosis has an insidious onset, diverse clinical manifestations, and is prone to misdiagnosis and missed diagnosis in clinical practice. The prognosis also has strong heterogeneity and is closely related to the extent of organ involvement at the time of diagnosis. In the past, the incidence of eye involvement in systemic AL amyloidosis patients was low, with various manifestations, only reported as case reports, and not regularly followed up with systemic treatment. Based on this, this project aims to assess the involvement of eyes and its appendages in patients with different stages of systemic light chain amyloidosis, with the goal of clarifying the ocular manifestations of this systemic disease and exploring early diagnostic indicators for the eye.

Primary Objective: To assess the involvement of the anterior segment of the eye, as well as the extraocular soft tissues and muscles, in patients with systemic light chain amyloidosis.

Secondary Objective: To assess the neuro-ophthalmic manifestations and changes in retinal choroidal blood flow in patients with systemic light chain amyloidosis.

Study Design: Observational study.

Study Population and Expected Enrollment: 80 patients with systemic light chain amyloidosis, 50 normal controls.

Study Duration: Six months of follow-up after the last subject is diagnosed and enrolled.

Intervention: Experimental Group: Patients with systemic light chain amyloidosis; Control Group: Subjects without systemic diseases.

ELIGIBILITY:
Case Group

Inclusion Criteria:

1. Patients diagnosed with "Systemic Light Chain Amyloidosis";
2. No other severe systemic underlying diseases that affect the examination;
3. Subjects voluntarily participate in this study, sign the informed consent form;
4. Age between 18-80 years old, no gender restrictions.

Exclusion Criteria:

1. Patients with eye diseases of clear causes such as ocular surface malignant tumors, corneal perforation, severe eye trauma, etc.;
2. Patients with nystagmus;
3. Severe ocular scar diseases; conjunctival scars with fornix shortening;
4. Current signs of infection, including fever and undergoing antibiotic treatment;
5. Mental abnormalities;
6. Pregnant or breastfeeding women, or women planning to become pregnant within 2 years;
7. NYHA Class IV: Heart disease patients cannot engage in any physical activity, with heart failure symptoms even at rest, and worsening with physical activity;
8. NT-proBNP > 8,500 ng/L.

Control Group

Inclusion Criteria:

1. Stable general condition, not patients with "Systemic Light Chain Amyloidosis";
2. No other severe systemic underlying diseases that affect the examination;
3. Subjects voluntarily participate in this study, sign the informed consent form;
4. Age between 18-80 years old, no gender restrictions.

Exclusion Criteria:

1. Patients with eye diseases of clear causes such as ocular surface malignant tumors, corneal perforation, severe eye trauma, etc.;
2. Patients with nystagmus;
3. Severe ocular scar diseases; conjunctival scars with fornix shortening;
4. Current signs of infection, including fever and undergoing antibiotic treatment;
5. Mental abnormalities;
6. Pregnant or breastfeeding women, or women planning to become pregnant within 2 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Source and Selection Method of Case Group: Patients diagnosed with "Systemic Light Chain Amyloidosis" or suspected of having "Systemic Light Chain Amyloidosis" and treated according to relevant diagnostic and treatment standards at tertiary hospitals. They are planned to undergo ocular screening at Zhongshan Ophthalmic Center of Sun Yat-sen University to exclude ocular and adnexal complications. It is expected that 80 cases of systemic light chain amyloidosis will participate in this study.
  Source and Selection Method of Control Group: Control group subjects are all sourced from the outpatient department of Zhongshan Ophthalmic Center of Sun Yat-sen University. It is expected that 50 cases of dry eye syndrome/cataract patients will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-08-13 (Estimated); Study Completion 2026-08-13 (Estimated)

PRIMARY OUTCOMES:
Conjunctival Mass | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Conjunctival Mass: The size of the yellowish-pink waxy mass on the bulbar or palpebral conjunctiva (if present, additional conjunctival confocal microscopy examination is performed to clarify the microscopic morphology of the mass).
Subconjunctival Hemorrhage Grading | Each system light chain amyloidosis patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Subconjunctival Hemorrhage: No conjunctival congestion is scored 0; mild diffuse conjunctival congestion is scored 1; moderate diffuse conjunctival congestion, with noticeable congestion near the fornices, is scored 2; severe diffuse conjunctival congestion with subconjunctival hemorrhage is scored 3.

SECONDARY OUTCOMES:
Periocular Purpura | Each system light chain amyloidosis patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Purple-red macules and papules on the skin around the orbit.
Ptosis | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Measure the degree to which the upper eyelid margin covers the cornea when both eyes are open and looking straight ahead. It is classified based on the degree of coverage: Mild: Coverage ≤4 mm, with a drooping amount of ≤2 mm; Moderate: Coverage >4～≤6 mm, drooping amount >2～≤4 mm; Severe: Coverage >6 mm, reaching the central part of the pupil, with a drooping amount >4 mm.
Vitreous Opacity | Each system light chain amyloidosis patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Fundus photography records the morphology of vitreous opacity, such as Weiss ring, flocculent, dense membranous, fine punctate, filamentous, reticular, etc.
Cup-to-Disc Ratio (C/D) | Each system light chain amyloidosis patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  After mydriasis (pupil > 6 mm), in a dark room, a skilled professional technician uses a digital fundus camera to adjust the machine's height, the subject's head position, and seating. The subject is instructed to open their eyes and focus on the cursor inside the machine, and two directional fundus photographs are taken for each eye (centered on the macula and the optic disc, respectively).
Visual Field | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  The extent of visual field defects is assessed according to the HPA (Humphrey Perimetry Analysis) international visual field staging method. An average deviation of <-6dB is considered mild, -6dB ≤ average deviation ≤ -12dB is moderate, and an average deviation >-12dB is severe.
Retinal Microvasculature | Each system light chain amyloidosis patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  OCTA measurement of superficial retinal vessel density in the foveal center (3mm)
Retinal Nerve Fiber Layer Thickness | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Heidelberg OCT measurement of retinal nerve fiber layer thickness in the foveal center (6mm)
Choroidal Thickness | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Heidelberg OCT measurement of choroidal thickness in the foveal center (6mm)
Cornea | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Corneal Dystrophy: Mucous drop dystrophy and lattice dystrophy of the cornea. If present, anterior segment OCT (Optical Coherence Tomography) is performed to assist in determining the depth of corneal opacity and deposition.
Visual Acuity | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  Uncorrected distant visual acuity is assessed using a Snellen chart. If the uncorrected distant visual acuity is less than 1.0, additional tests including computerized refraction and corrected distant visual acuity are performed.
Non-contact Intraocular Pressure | Each patient will be followed up once every 2 months, for a total of 4 follow-ups, over a 6-month period, to observe any ocular complications and progression.
  The tonometer measures the intraocular pressure and displays the result on the screen, taking three consecutive measurements. If an erroneous value is detected, the subject rests and adjusts for 1 minute before repeating the intraocular pressure measurement three times to record the accurate data.

CONTACTS AND LOCATIONS:
Overall Officials: chang he, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China